CLINICAL TRIAL: NCT04560517
Title: Study of Remission Factors in Anorexia Nervosa of Adult Women (REMANO)
Brief Title: Remission Factors in Anorexia Nervosa
Acronym: REMANO
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C18-39; 2019-A01352-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-08-25; First posted 2020-09-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: eating disorder; anorexia nervosa; delay discounting; ghrelin; genetic; epigenetic
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group of patients suffering from anorexia nervosa: Are considered, all patients admitted to the Hospitalization unit for eating disorders of the Mental Health and Brain Disorders Clinic
- Group of healthy volonteers: The control volunteers are recruited by posting within various institutions of the Paris Descartes faculty. Participants themselves contact the clinical research nurse, whose number is clearly stated on the poster.

SUMMARY:
Anorexia Nervosa (AN) is a complex and multifactorial psychiatric disease that affects mostly women and is characterized by a self-restriction of food intake leading to life-threatening consequences whose underlying mechanisms are largely unexplored. AN encompasses a constellation of risk factors including genetic, biological, neuro-psychological and social factors. Although AN has a prevalence of only 1-3% in the general population, it has the highest mortality rate amongst any psychiatric disorder. Recovery of normal feeding behaviour in patients often requires several months with a large between-patient variability and a high percentage of relapse, which can occur in 35 to 41% of the patients. There is a huge unmet need for optimal understanding of processes underlying relapse. Reward processing abnormalities represents an important hypothesis underlying AN development and perpetuation. We aim to investigate the mechanisms that contribute to the maintenance and chronicity of the disease after inpatient treatment with a longitudinal design across intensive standardized inpatient treatment. We will challenge our hypothesis through brain imaging, neuropsychological, metabolic and genetic approaches. One hundred twenty-five AN female patients admitted for intensive inpatient treatment will be recruited and evaluated: at admission, after weight recovery and at 6 months after discharge with neurocognitive tests (including the Delay Discounting Task), genetic/epigenetic examination, hormonal blood samples (at each visit and repeated sampling around a meal for a 10-patient subgroup) and brain imaging (including fMRI during a Delay Discounting Task for fifty patients). One hundred healthy controls will be also recruited and be subjected to the same study procedures.

ELIGIBILITY:
Inclusion Criteria:

* DMS 5 criteria for Anorexia Nervosa
* BMI < 18.5 kg/m²
* Being able to consent
* fluent in French
* Being affiliated to a social security scheme or being the beneficiary of such a scheme.
* Having signed the informed consent

Exclusion Criteria:

* Deprived of liberty subject (judicial or administrative decision)
* Refusal to participate
* Presenting an unstabilized serious physical illness or psychiatric disorder compromising the follow up according investigator evaluation
* Contraindication for IRMf
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients :
  all female patients integrating inpatient treatment program for Anorexia Nervosa at the Clinique des Maladies Mentales et de l'Encéphale in Paris, France
  Control group :
  Female aged from 18 to 65 years old without any psychiatric disorder
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Delay Discounting Task score after weight recovery | after complete weight recovery (4+/-2 months after inclusion)
  Comparaison of this score to remission status six months post discharge

SECONDARY OUTCOMES:
Delay Discounting Task score after weight recovery compared to control | after weight recovery (4+/-2 months after baseline)
Bold signal difference during Delay Discounting Task in fMRI | Baseline (M0) and after weight recovery for patient (4+/-2 months after baseline) ; Baseline and 4 months later for healthy controls
Evolution of brain volums in MRI | Baseline (M0), after weight recovery (4+/-2 months after baseline)
Evolution of fronto striatal connectivity in MRI | Baseline (M0), after weight recovery (4+/-2 months after baseline)
Evolution of total, acyl and desacyl ghrelin plasma level | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
Evolution of total, acyl and desacyl ghrelin plasma level around a meal | Baseline (Month 0), after weight recovery (4+/-2 months after baseline) during meal
Exome analysis | Baseline (M0)
Evolution of BDNF gene methylation | Baseline (M0), after weight recovery (4+/-2 months after baseline)
Evolution of EDI-2 score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of eating disorder dimensions during weight recovery predicting relapse
Evolution of EAI score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of physical activity addiction during weight recovery predicting relapse
Evolution of GLT score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of the level of physical activity during weight recovery predicting relapse
Evolution of YBS score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of obession and compulsion during weight recovery predicting relapse
Evolution of HADS score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of anxiety and depression during weight recovery predicting relapse
Evolution of Brixton score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of neuropsychological performance during weight recovery predicting relapse
Evolution of TMT score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of neuropsychological performance during weight recovery predicting relapse
Evolution of Slips of action neurocognitive score | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of neuropsychological performance during weight recovery predicting relapse
Evolution of pupillometry to social, food and body image pictures | Baseline (M0), after weight recovery (4+/-2 months after baseline) and 6 months post discharge
  Evaluate the evolution of neuropsychological performance during weight recovery predicting relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier St Anne, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duriez P, Tolle V, Ramoz N, Kimmel E, Charron S, Viltart O, Lebrun N, Bienvenu T, Fadigas M, Oppenheim C, Gorwood P. Assessing biomarkers of remission in female patients with anorexia nervosa (REMANO): a protocol for a prospective cohort study with a nested case-control study using clinical, neurocognitive, biological, genetic, epigenetic and neuroimaging markers in a French specialised inpatient unit. BMJ Open. 2024 Jun 25;14(6):e077260. doi: 10.1136/bmjopen-2023-077260. PMID 38925688